CLINICAL TRIAL: NCT00745095
Title: Efficacy and Safety of Bowel Preparations for Colonoscopy in SCI
Brief Title: Efficacy and Safety of Standard Oral Colonoscopic Preparations With or Without Neostigmine Compared to Pulse-Irrigation Colonic Lavage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: A6428-R; KOR-09-10 (Other: James J. Peters VA Medical Center)
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-05

CONDITIONS: Spinal Cord Injury
Keywords: Safety; Efficacy; Colonoscopy; PIEE; MoviPrep; Neostigmine; Glycopyrrolate
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SCI MoviPrep® (without NG) (No Intervention): (Spinal Cord Injury (SCI), glomerular filtration rate (GFR)<=50ml/min and SCI, GFR>=50ml/min) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid [MoviPrep®] (without neostigmine plus glycopyrrolate [NG])
- SCI PIEE (without NG) (No Intervention): (Spinal Cord Injury (SCI), glomerular filtration rate (GFR)>=50ml/min) pulsed irrigation enhanced evacuation [PIEE] (without neostigmine plus glycopyrrolate [NG])
- Control MoviPrep® only (No Intervention): (Control, glomerular filtration rate (GFR)>=50ml/min) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid (MoviPrep®) only (no NG)
- Control PIEE only (No Intervention): (Control, glomerular filtration rate (GFR)>=50ml/min), pulsed irrigation enhanced evacuation (PIEE) only (no NG)
- SCI MoviPrep® (with NG) (Experimental): (Spinal Cord Injury (SCI), glomerular filtration rate (GFR)<=50ml/min and SCI GFR>=50ml/min) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid [MoviPrep®] (with neostigmine plus glycopyrrolate [NG])
  Interventions: Drug: Neostigmine
- SCI PIEE (with NG) (Experimental): (Spinal Cord Injury (SCI), glomerular filtration rate (GFR)>=50ml/min) pulsed irrigation enhanced evacuation (PIEE) (with neostigmine plus glycopyrrolate [NG])
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Neostigmine — Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
  Arms: SCI MoviPrep® (with NG); SCI PIEE (with NG)

SUMMARY:
The annual incidence of colorectal cancer in the US during 2005 was approximately 150,000 cases and this neoplasm claimed 56,000 lives (American Cancer Society). Detection (and removal) of colonic polyps is now the central strategy in reducing the risk of colon cancer. Thus, failure to detect and remove small cancers and polyps can have dire consequences. Although it has not been shown that persons with spinal cord injury (SCI) have an increased risk of this disease, there is no reason to assume that the incidence after SCI would be less than that of the general population.

Colonoscopy would appear to be a better approach to colon cancer screening after SCI but may also be unreliable if bowel evacuation is unsatisfactory for complete large bowel visualization. Poor colonoscopic visualization is a major concern in persons with SCI because they have long-standing difficulty with evacuation (DWE) and might not respond in a predictable or satisfactory manner to the conventional bowel preparations used for colonoscopy. Furthermore, to the extent that bowel preparation for colonoscopy is unsatisfactory in persons with SCI, the putative benefits of colonoscopy in reducing colon cancer mortality may not be realized.

In the absence of effective regimens for bowel preparation in persons with SCI, we suspect that the documented benefits of screening colonoscopy in the able-bodied may not generalize to persons with SCI. Regardless, these observations support the need for improved bowel preparation approaches in persons with SCI. One such approach might involve the adjunctive administration of prokinetic drugs to standard practices. A prokinetic agent that might be beneficial in this context is neostigmine, an anticholinesterase inhibitor with prominent parasympathomimetic actions (stimulation of peristalsis) on the colon. We have studied neostigmine extensively in persons with SCI and have shown that, when given in combination with glycopyrrolate, this approach to stimulate bowel evacuation is safe and effective for bowel evacuation.

DETAILED DESCRIPTION:
The annual incidence of colorectal cancer in the US during 2005 was approximately 150,000 cases and this neoplasm claimed 56,000 lives (American Cancer Society). Detection (and removal) of colonic polyps is now the central strategy in reducing the risk of colon cancer. Thus, failure to detect and remove small cancers and polyps can have dire consequences. Although it has not been shown that persons with spinal cord injury (SCI) have an increased risk of this disease, there is no reason to assume that the incidence after SCI would be less than that of the general population.

Colonoscopy would appear to be a better approach to colon cancer screening after SCI but may also be unreliable if bowel evacuation is unsatisfactory for complete large bowel visualization. Poor colonoscopic visualization is a major concern in persons with SCI because they have long-standing difficulty with evacuation (DWE) and might not respond in a predictable or satisfactory manner to the conventional bowel preparations used for colonoscopy. Furthermore, to the extent that bowel preparation for colonoscopy is unsatisfactory in persons with SCI, the putative benefits of colonoscopy in reducing colon cancer mortality may not be realized.

In the absence of effective regimens for bowel preparation in persons with SCI, we suspect that the documented benefits of screening colonoscopy in the able-bodied may not generalize to persons with SCI. Regardless, these observations support the need for improved bowel preparation approaches in persons with SCI. One such approach might involve the adjunctive administration of prokinetic drugs to standard practices. A prokinetic agent that might be beneficial in this context is neostigmine, an anticholinesterase inhibitor with prominent parasympathomimetic actions (stimulation of peristalsis) on the colon. We have studied neostigmine extensively in persons with SCI and have shown that, when given in combination with glycopyrrolate, this approach to stimulate bowel evacuation is safe and effective for bowel evacuation.

ELIGIBILITY:
Inclusion Criteria:

1. SCI and able-bodied patients with clinical indication for a colonoscopic examination

Exclusion Criteria:

1. Able-bodied patients with a GFR 50ml/min.
2. SCI and able-bodied patients who are not candidates for elective colonoscopy (i.e., those with recent myocardial infarction, terminal illness, etc.)
3. SCI and able-bodied patients who have a contraindication to PEG and/or ascorbic acid administration (i.e., those with colonic obstruction, etc.)
4. SCI and able-bodied patients who have a contraindication for magnesium citrate (i.e., those with poor renal function, class 2 or greater symptomatic heart failure, ascites)
5. SCI and able-bodied patients with a history of bradyarrhythmia, active coronary artery disease or asthma will also be excluded from receiving neostigmine/glycopyrrolate
6. Known hypersensitivity to neostigmine or glycopyrrolate
7. Potential for pregnancy. Women who are sexually active and of childbearing potential (i.e. not surgically sterile or at least 2 years postmenopausal) must have negative serum pregnancy test.)
8. Lactating/nursing females
9. SCI patients with known adverse reactions to per-rectal colonic lavage.
10. SCI patients with a serum sodium <130 mM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Korsten, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Derived] Lyons BL, Korsten MA, Spungen AM, Radulovic M, Rosman AS, Hunt K, Galea MD, Kornfeld SD, Yen C, Bauman WA. Comparison between pulsed irrigation enhanced evacuation and polyethylene glycol-electrolyte lavage solution for bowel preparation prior to elective colonoscopy in veterans with spinal cord injury. J Spinal Cord Med. 2015 Nov;38(6):805-11. doi: 10.1179/2045772314Y.0000000256. Epub 2014 Aug 6. PMID 25096918

RESULTS

PARTICIPANT FLOW:
Groups:
- SCI MoviPrep® (Without NG): (Spinal Cord Injury [SCI], glomerular filtration rate [GFR]<=50 and SCI, GFR>=50) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid [MoviPrep®] (without neostigmine plus glycopyrrolate [NG])
- SCI MoviPrep® (With NG): (Spinal Cord Injury [SCI], glomerular filtration rate [GFR]<=50ml/min and SCI, GFR>=50ml/min) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid [MoviPrep®] (with neostigmine plus glycopyrrolate [NG])
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- SCI PIEE (Without NG): (Spinal Cord Injury [SCI], glomerular filtration rate [GFR]>=50ml/min) pulsed irrigation enhanced evacuation (PIEE) (without neostigmine plus glycopyrrolate [NG])
- SCI PIEE (With NG): (Spinal Cord Injury [SCI], glomerular filtration rate [GFR]>=50ml/min) pulsed irrigation enhanced evacuation (PIEE) (with neostigmine plus glycopyrrolate [NG])
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- Control MoviPrep® Only: (Control, GFR>=50ml/min) low-volume polyethylene glycol-electrolyte lavage with ascorbic acid [MoviPrep®] only (no neostigmine plus glycopyrrolate [NG])
- Control PIEE Only: (Control, GFR>=50ml/min) PIEE only (no neostigmine plus glycopyrrolate [NG])
Period: Overall Study
Arm/Group | SCI MoviPrep® (Without NG) | SCI MoviPrep® (With NG) | SCI PIEE (Without NG) | SCI PIEE (With NG) | Control MoviPrep® Only | Control PIEE Only
Started | 15 | 15 | 15 | 15 | 150 | 150
Completed | 14 | 13 | 12 | 12 | 28 | 27
Not Completed | 1 | 2 | 3 | 3 | 122 | 123
Not completed — Declined to participate | 1 | 0 | 0 | 0 | 92 | 95
Not completed — Ineligible due to GFR criteria | 0 | 2 | 3 | 3 | 30 | 28

BASELINE CHARACTERISTICS:
Groups:
- SCI MoviPrep® (Without NG): (SCI, GFR<=50ml/min and GFR>=50ml/min) MoviPrep® (without NG)
- SCI MoviPrep® (With NG): (SCI, GFR<=50ml/min and GFR>=50ml/min) MoviPrep® (without NG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- SCI PIEE (Without NG): (SCI, GFR>=50ml/min) PIEE ( without NG)
- SCI PIEE (With NG): (SCI, GFR>=50ml/min) PIEE (with NG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- Control MoviPrep® Only: (Control, GFR>=50ml/min) MoviPrep® only (no NG)
- Control PIEE Only: (Control, GFR>=50ml/min) PIEE only (no NG)
- Total: Total of all reporting groups
Arm/Group | SCI MoviPrep® (Without NG) | SCI MoviPrep® (With NG) | SCI PIEE (Without NG) | SCI PIEE (With NG) | Control MoviPrep® Only | Control PIEE Only | Total
Number analyzed (Participants) | 14 | 13 | 12 | 12 | 28 | 27 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8) | 65 (6) | 61 (11) | 58 (5) | 58 (10) | 60 (9) | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2 | 2 | 6
  Male | 14 | 13 | 11 | 11 | 26 | 25 | 100
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 12 | 12 | 28 | 27 | 106

OUTCOME MEASURES:

1. Primary Outcome: Quality of Bowel Preparation
Description: The quality of bowel preparation was determined by using the Ottawa Scale for bowel Evacuation. The range of this score is from 0 (perfectly clean and dry colon) to 14 ( a colon filled with stool and liquid). The right, mid and rectosigmoid colon were independently rated from 0-4 and fluid quality of entire colon was recorded with an additional score of 0-2. The total Ottawa Score is calculated by the sum of the independent scores of all three sections of the colon plus the fluid content.
Time Frame: 1-2 days following intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SCI MoviPrep® (Without NG): (SCI, GFR<=50 and GFR >=50) MoviPrep® (without NG)
- SCI MoviPrep® (With NG): (SCI, GFR<=50ml/min and GFR >=50ml/min) MoviPrep® (withNG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- SCI PIEE (Without NG): (SCI, GFR>=50ml/min) PIEE (without NG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
Arm/Group | SCI MoviPrep® (Without NG) | SCI MoviPrep® (With NG) | SCI PIEE (Without NG) | SCI PIEE (With NG) | Control MoviPrep® Only | Control PIEE Only
Number analyzed (Participants) | 14 | 13 | 12 | 12 | 28 | 27
units on a scale | 3.4 (1.6) | 2.5 (2.4) | 3.6 (3.1) | 7.4 (5.0) | 1.8 (1.9) | 6.9 (4.8)

2. Secondary Outcome: Polyp Detection
Description: The number of polyps detected during colonoscopic procedures were recorded and compared to each bowel cleansing preparation.
Time Frame: Time of Study
Measure: Mean (Standard Deviation); unit: Number of polyps detected (numerical)
Groups:
- SCI MoviPrep® (Without NG): (SCI, GFR<=50ml/min and GFR >=50ml/min) MoviPrep® ( without NG)
- SCI MoviPrep® (With NG): (SCI, GFR<=50ml/min and GFR >=50ml/min) MoviPrep® (with NG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- SCI PIEE ( Without NG): (SCI, GFR>=50ml/min) PIEE ( without NG)
Arm/Group | SCI MoviPrep® (Without NG) | SCI MoviPrep® (With NG) | SCI PIEE ( Without NG) | SCI PIEE (With NG) | Control MoviPrep® Only | Control PIEE Only
Number analyzed (Participants) | 14 | 13 | 12 | 12 | 28 | 27
Number of polyps detected (numerical) | 1.3 (1.7) | 1.3 (1.5) | 0.4 (1.2) | 0.5 (1.2) | 0.9 (1.0) | 0.3 (0.8)

ADVERSE EVENTS:
Groups:
- SCI MoviPrep® (Without NG): (SCI, GFR<=50ml/min and GFR >=50ml/min) MoviPrep (without NG)
- SCI MoviPrep® (With NG): (SCI, GFR<=50ml/min and GFR >=50ml/min) MoviPrep (with NG)
  Neostigmine: Neostigmine will be administered in 20, 40, and 60mg doses until an individualized dose-response relationship is established
- SCI PIEE Only: (Control, GFR>=50ml/min) PIEE only (no NG)
Arm/Group | SCI MoviPrep® (Without NG) | SCI MoviPrep® (With NG) | SCI PIEE (Without NG) | SCI PIEE (With NG) | Control MoviPrep® Only | SCI PIEE Only
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12 | 0/12 | 1/28 | 1/27
Other Adverse Events (participants affected / at risk) | 1/14 | 7/13 | 4/12 | 10/12 | 4/28 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SCI MoviPrep® (Without NG) (N=14) | SCI MoviPrep® (With NG) (N=13) | SCI PIEE (Without NG) (N=12) | SCI PIEE (With NG) (N=12) | Control MoviPrep® Only (N=28) | SCI PIEE Only (N=27)
Death (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 — This account was unrelated to study participation since the subject passed away years after their completion. However since the subject passed away while the the study was open, this event was recorded.
Renal Problems (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Possibly related to the subject's participation in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCI MoviPrep® (Without NG) (N=14) | SCI MoviPrep® (With NG) (N=13) | SCI PIEE (Without NG) (N=12) | SCI PIEE (With NG) (N=12) | Control MoviPrep® Only (N=28) | SCI PIEE Only (N=27)
Orthostatic Hypotension (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
GI discomfort, bloating, distention (Gastrointestinal disorders) | 1 | 7 | 3 | 7 | 4 | 13 — Symptoms reported by patients during study participation
Unable to complete preparation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 | 0 | 7 — Patients who were unable to successfully have a proper and complete bowel evacuation prior to colonoscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes